CLINICAL TRIAL: NCT06090370
Title: Reducing Silica Exposure Among Brick Kiln Workers in Nepal: A Human-centered Design Framework to Develop a Personal Protective Equipment Training Intervention
Brief Title: Reducing Silica Exposure Among Brick Kiln Workers in Nepal
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Tribhuvan University (Unknown); Chiesi Foundation (Unknown); National Institutes of Health (NIH) (NIH); Duke University (Other); Fogarty International Center of the National Institute of Health (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00387104; D43TW009340 (NIH)
Record Dates: First submitted 2023-10-12; First posted 2023-10-19 (Actual); Last update posted 2024-06-24 (Actual); Status verified 2024-06

CONDITIONS: Silicosis
Keywords: Silica Exposure; Brick Kiln; Personal Protective Equipment (PPE) Program
MeSH Terms: conditions — Silicosis | interventions — N95 Respirators; Surveys and Questionnaires

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Baseline Survey: Silicosis and Personal Protective Equipment (Experimental)
  Interventions: Other: Baseline Survey
- Design of Personal Protective Equipment Training Workshop (Experimental)
  Interventions: Other: Design of Workshop
- Pilot Study: Personal Protective Equipment Training Program (Experimental): A small training program will be offered to brick kiln workers to determine preferred PPE type, feasibility in the work environment and proper usage of PPE.
  Interventions: Device: N95 Respirator; Device: Protective Eyewear
- Feedback Workshop on Pilot Personal Protective Equipment Training Program (Experimental)
  Interventions: Other: Training Workshop Pilot

INTERVENTIONS:
Device: N95 Respirator — The participants in this group will be provided with N95 respirator masks to protect from dust and debris while working in the brick kiln and trained on proper usage.
  Arms: Pilot Study: Personal Protective Equipment Training Program
Device: Protective Eyewear — The participants in this group will be provided with eye wear to protect the eyes from dust and debris while working in the brick kiln and trained on proper usage
  Arms: Pilot Study: Personal Protective Equipment Training Program
Other: Baseline Survey — A quantitative, cross-sectional survey will be distributed to enrolled participants to understand baseline worker perceptions on silicosis and personal protective equipment (PPE).
  Arms: Baseline Survey: Silicosis and Personal Protective Equipment
Other: Design of Workshop — A co-creation human centered design workshop to elicit feedback on PPE training prototypes and types of PPE.
  Arms: Design of Personal Protective Equipment Training Workshop
Other: Training Workshop Pilot — Qualitative workshops will be held to elicit feedback on the piloted PPE training program.
  Arms: Feedback Workshop on Pilot Personal Protective Equipment Training Program

SUMMARY:
Inhaling respirable silica increases the risk for silicosis, an incurable and debilitating lung disease. In South Asia, one high-risk industry is brick manufacturing, where more than 4 million manual laborers mold bricks by hand. In Nepal, brick manufacturing employs over 200,000 workers across 1,200 registered brick kilns. These workers are exposed to respirable silica concentrations 1.4 to 6.6 times higher than the limits set by the U.S. National Institute for Occupational Safety and Health. Preventing silicosis is paramount, as the average brick kiln worker cannot afford medical care and only 6.8% receive regular health checks. Few studies have evaluated interventions in brick kiln workers to reduce silica exposure and prevent silicosis.

One promising intervention involves providing workers who are exposed to silica above the permissible exposure limit with personal protective equipment (PPE), specifically respirators. When properly used, respirators decrease silica inhalation and the risk of silicosis. Brick kiln workers in Nepal do not use any PPE. Several studies have explored PPE barriers and have evaluated the feasibility of implementing PPE but to date none have been conducted in Nepali brick kiln workers. To close this gap, the goal of this research is a human-centered design approach to develop and pilot a PPE training program in one brick kiln in Nepal guided by the Discover, Design, Build, and Test (DDBT) framework.

This research is necessary to understand the Nepali context and to efficiently develop appropriate and feasible PPE intervention components that will be trialed in future research.

DETAILED DESCRIPTION:
Workers will be recruited from Bhaktapur, a district in the Kathmandu Valley.

The investigators will conduct a four-part study. Part 1 will involve a quantitative, cross-sectional survey to understand baseline worker perceptions on silicosis and personal protective equipment (PPE). Part 2 will comprise qualitative co-creation human-centered design workshops to elicit feedback on PPE training prototypes and types of PPE. Part 3 will be a small feasibility pilot of the training program and most preferred type of PPE. Part 4 will comprise qualitative workshops to elicit feedback on the piloted PPE training program.

The same participants may participate in Part 1 and 2. Participants in Part 3 will be a distinct group from those who participated in Parts 1 and 2.

Assessments will include:

Aim 1: Characterize knowledge gaps and behaviors influencing PPE use among brick kiln workers in Bhaktapur, Nepal Method: Quantitative, cross-sectional survey to understand baseline worker perceptions on silicosis and personal protective equipment (PPE). N = 100 workers.

Aim 2: Design a personal protective equipment (PPE) training program for brick kiln workers in Nepal through a human-centered design approach Method: 4 qualitative co-creation human-centered design workshops. N = 20 - 40 workers.

Aim 3: Evaluate acceptability, appropriateness, and feasibility of personal protective equipment (PPE) training through a pilot among brick kiln workers in Nepal Method: Feasibility pilot study at 1 brick kiln for 3 weeks. N = 20 workers (intervention) and N = 20 workers (control). 3 qualitative co-creation human-centered design workshops to elicit feedback after the pilot. N = 10 - 20 workers.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Active Brick Kiln Workers in Bhaktapur, Nepal
* Cognitively capable to provide informed consent

Exclusion Criteria:

* Less than 18 years old
* Non Brick Kiln Workers
* Not cognitively capable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2024-01-24 (Actual); Primary Completion 2024-06-20 (Actual); Study Completion 2024-06-20 (Actual)

PRIMARY OUTCOMES:
Feasibility as assessed by The Feasibility of Intervention Measure (FIM) score | 12 months
  Feasibility will be measured using the Feasibility of Intervention Measure which includes 4 questions with 5-point likert response options, Completely disagree (1) - Completely agree (5). Higher score, higher agreement of feasibility.

CONTACTS AND LOCATIONS:
Overall Officials: William Checkley, MD, PhD, Principal Investigator — Johns Hopkins School of Medicine
Locations (3):
- United States (2):
  - Johns Hopkins University, Baltimore, Maryland
  - Duke University, Durham, North Carolina
- Tribhuvan University, Maharajgunj, Kathmandu, Nepal